CLINICAL TRIAL: NCT03876912
Title: The Effect of Androgen Deprivation Therapy on the Expression of Prostate Specific Membrane Antigen (PSMA) Evaluated With 18F-PSMA PET/CT in Treatment naïve Metastatic Prostate Cancer Patients
Brief Title: The Effect of ADT on PSMA Expression in Metastatic Prostate Cancer
Acronym: ADTPSMA2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADTPSMA2
Record Dates: First submitted 2019-03-14; First posted 2019-03-15 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Specific Membrane Antigen; GnRH antagonist; Positron Emission Tomography; PSMA-PET/CT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GnRH antagonist (Experimental): Administration of GnRH antagonist (subcutaneous injection, 240 mg) after baseline 18F-PSMA 1007 PET/CT.Then 18F-PSMA 1007 PET/CT is repeated 3 weeks after ADT and at development of CRPC
  Interventions: Drug: GnRH antagonist

INTERVENTIONS:
Drug: GnRH antagonist — 18F-PSMA 1007 PET/CT before, 3 weeks after ADT, at 1 year and at CRPC in 35 patients. 18F-FDG PET/CT in a subgroup of 20 patients before ADT.
  Other Names: Degarelix

SUMMARY:
Thirty-five men with newly diagnosed, metastatic prostate cancer are scanned with 18F-PSMA 1007 PET/CT at baseline, 3 weeks after the initiation of GnRH-antagonist, at one year and at the time of castration resistant prostate cancer (CRPC). The aim of the study is to classify metastatic lesions into those with PSMA-flare and those without and determine their potential to progress during the follow-up until CRPC.

DETAILED DESCRIPTION:
In metastatic prostate cancer androgen deprivation therapy (ADT) has been traditionally used as a first line approach. Based on histological studies, animal models and PSMA-PET imaging, it is known that administration of ADT increases prostate specific membrane antigen (PSMA) expression.

Preliminary results of our previous prospective clinical trial (clinicaltrials.gov identifier: NCT03313726) with nine men demonstrated a heterogenous flare in PSMA expression 2-3 weeks after ADT, more evidently in bone metastases. Our hypothesis is that metastatic lesions having PSMA-flare respond differently to ADT and have different outcome than those without PSMA-flare. Therefore, the objective of the study is to demonstrate the PSMA-flare seen in bone lesions 3 weeks after ADT and then determine the potential predictive value of the phenomenon in the progression to castration resistant prostate cancer (CRPC).

Thirty-five men with newly diagnosed, metastatic PC will undergo 18F-PSMA 1007 PET/CT before and 3 weeks after the initiation of sub-cutaneous injection of GnRH-antagonist (Degarelix, Firmagon®). A subgroup of 20 patients will receive an additional FDG PET/CT scan before ADT to investigate whether lesions with PSMA flare show a different metabolic behaviour on FDG PET. During the follow-up, 18F-PSMA 1007 PET/CT will be also performed once a year. Finally all patients will repeat 18F-PSMA 1007 PET/CT at the time of CRPC. In addition to imaging, PSA is measured, and blood drawn for androgen levels and biomarkers in three months interval.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 to 85 years old
* Language spoken: Finnish
* Diagnosis: Histologically confirmed adenocarcinoma of prostate
* Adequate histological sampling consisting of at least 3 biopsy samples from each lobe
* No previous surgical, radiation or endocrine treatment for prostate carcinoma
* Clinical stage:T1c-T4NanyM1
* Serum creatinine ≤ 1,5 x ULN
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethical Committee approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* Previous PC treatment
* Uncontrolled serious infection
* Prior usage of 5-ARI medication in past 12 months

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer patients
Enrollment: 35 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
PSMA-flare after ADT | 2-3 weeks
  Comparison of mean increase of SUVmax in 18F-PSMA 1007 PET between bone lesions and prostatic lesions after the initiation of ADT

SECONDARY OUTCOMES:
PSMA-flare in the follow-up until CRPC | 2-3 years
  Compare SUVmax of lesions with PSMA flare and those without during the follow-up and at CRPC

CONTACTS AND LOCATIONS:
Overall Officials: Jukka Kemppainen, Adj.Prof., Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Malaspina S, Ettala O, Tolvanen T, Rajander J, Eskola O, Bostrom PJ, Kemppainen J. Flare on [18F]PSMA-1007 PET/CT after short-term androgen deprivation therapy and its correlation to FDG uptake: possible marker of tumor aggressiveness in treatment-naive metastatic prostate cancer patients. Eur J Nucl Med Mol Imaging. 2023 Jan;50(2):613-621. doi: 10.1007/s00259-022-05970-y. Epub 2022 Sep 26. PMID 36161511